CLINICAL TRIAL: NCT03563560
Title: A Phase 1 Clinical Study of DSP-2033 (Alvocidib) in Combination With Cytarabine/Mitoxantrone or Cytarabine/Daunorubicin (7+3) in Patients With Acute Myeloid Leukemia
Brief Title: A Study of DSP-2033 (Alvocidib) in Patients With Acute Myeloid Leukemia
Acronym: AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC850101
Record Dates: First submitted 2018-03-21; First posted 2018-06-20 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Newly diagnosed AML; Relapsed/refractory AML; Alvocidib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — alvocidib; Cytarabine; Mitoxantrone; Daunorubicin

STUDY DESIGN:
Intervention Model Description: This study consists of 2 cohorts of the ACM regimen part and 1 cohort of the A+7+3 regimen part.
Masking Description: Open labeled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACM regimen (Experimental): ACM regimen is for Japanese patients with relapsed or refractory AML.
  Interventions: Drug: Alvocidib; Drug: Cytarabine; Drug: Mitoxantrone
- A+7+3 regimen (Experimental): A+7+3 regimen is for Japanese newly diagnosed AML patients.
  Interventions: Drug: Alvocidib; Drug: Cytarabine; Drug: Daunorubicine

INTERVENTIONS:
Drug: Alvocidib — ACM regimen:30 mg/60 mg, 30-minute intravenous (IV) infusion, followed 4-hour IV infusion from Day 1 to Day 3 A+7+3 regimen: recommended dose (RD), 30-minute IV infusion, followed 4-hour IV infusion from Day 1 to Day 3
  Other Names: DSP-2033
Drug: Cytarabine — 300 or 667 mg/m2/day, 72-hour continuous IV infusion starting on Day 6 (ACM regimen)
  Other Names: DSP-AraC
  Arms: ACM regimen
Drug: Mitoxantrone — 14 or 40 mg/m2/day, IV infusion over 1 hour to 2 hours at 12 hours after the end of DSP-AraC administration (acceptable range + 3 hours)
  Other Names: DSP-MIT
  Arms: ACM regimen
Drug: Cytarabine — 100 mg/m2/day, continuous IV infusion for 7 days from Day 5 to Day 11 (A+7+3 regimen)
  Arms: A+7+3 regimen
Drug: Daunorubicine — 60 mg/m2/day, 30-minute IV infusion for 3 days from Day 5 to Day 7
  Other Names: DSP-DNR
  Arms: A+7+3 regimen

SUMMARY:
This is an open label, multi-center, phase 1 study of DSP-2033 (Alvocidib) in combination with cytarabine/mitoxantrone (ACM regimen) or cytarabine/daunorubicin (A+7+3 regimen) in patients with acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
This study consists of 2 cohorts of the ACM regimen part for Japanese relapsed/refractory AML patients and 1 cohort of the A+7+3 regimen part for Japanese newly diagnosed AML patients. The purpose of this study are as below.

1. To evaluate the safety of DSP-2033 (Alvocidib) in combination with cytarabine/mitoxantrone (ACM regimen) in Japanese patients with relapsed or refractory AML and to confirm its tolerability.
2. To evaluate the safety of DSP-2033 （Alvocidib) in combination with cytarabine/daunorubicin (A+7+3 regimen) in Japanese newly diagnosed AML patients and to confirm its tolerability.

ELIGIBILITY:
Inclusion Criteria:

[For all parts]

1. Japanese patients diagnosed with AML by the 4th edition of WHO criteria.
2. Patients aged between 20 and 64 at acquisition of informed consent.
3. Have received an adequate explanation of the objectives/contents of the clinical study, anticipated therapeutic effects/pharmacology, and risks to his/her understanding, and voluntarily provide written informed consent to participation in the clinical study.
4. Have an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2 at entry.
5. Have a left ventricular ejection fraction (LVEF) ≥ 50% determined by echocardiography or multigated acquisition (MUGA) scan within 14 days prior to entry.
6. Have an arterial oxygen saturation (SpO2) ≥ 90% within 14 days prior to entry.
7. The laboratory test within 14 days prior to entry (for multiple tests, the most recent before the entry) meet the following criteria for major organ function.

   1. Serum creatinine ≤ 1.5 x the upper limit of normal (ULN) of the institutional reference standard
   2. AST and ALT ≤ 2 x ULN of the institutional reference standard
   3. Total bilirubin ≤ 2.0 mg/dL
8. Female patients of childbearing potential must have negative pregnancy test results at entry.
9. Female patients or patients with partners of childbearing potential must agree to use an appropriate method of contraception for a period between acquisition of informed consent and 6 months (180 days) after the final dose so that patients or female partners would not become pregnant.

   [ACM regimen part] In addition to the inclusion criteria for all parts, patients must meet the following criterion.
10. AML patients who could not attain remission after 1 or 2 cycles of potent chemotherapy with anthracycline, cytarabine, and etoposide, or potent chemotherapy with anthracycline and cytarabine. Or patients with 1st or 2nd recurrent AML after complete remission following initial therapy.

    [A+7+3 regimen part] In addition to the inclusion criteria for all parts, patients must meet the following criterion
11. Treatment naive AML patients.

Exclusion Criteria:

[For all parts]

1. Diagnosed with acute promyelocytic leukemia (APL) (FAB classification: M3).
2. Received a transplantation such as hematopoietic stem cell transplant.
3. Have active central nervous system (CNS) leukemia.
4. Complicated by ≥ Grade 3 infection as specified in Common Terminology Criteria for Adverse Events version 4.03 (CTCAE v4.03).
5. HIV antibody, HBs antigen, or HCV antibody tested positive within 90 days prior to entry.
6. Have New York Heart Association (NYHA) cardiac function classification III or IV heart disease or a history, ≥ Grade 3 arrhythmia, angina pectoris or abnormal electrocardiogram (ECG) findings as specified in CTCAE v4.03 or a history of these above.
7. Have a disease that may interfere with the study treatment, such as interstitial pneumonia, pulmonary fibrosis, or active tuberculosis.
8. Complicated by uncontrolled disseminated intravascular coagulation.
9. Have other active malignancies (synchronous multiple malignancies and metachronous multiple malignancies with a disease-free interval not more than 5 years. However, carcinoma in situ that is determined to be cured by local treatment or lesions equivalent to mucosal carcinoma are not included in active multiple malignancies.)
10. Have an uncontrolled complication.
11. Complicated by mental deficits or have a history of mental deficits. However, patients who are able to comply with the study protocol can be included at the discretion of a physician.
12. Complicated by varicella.
13. Received any previous treatment with DSP-2033 or other CDK inhibitors.
14. Received any investigational product or post-marketing clinical study drug within 3 months (90 days) prior to entry.
15. Pregnant or lactating women*)

    *) If a lactating woman agrees to discontinue breast feeding between acquisition of informed consent and 6 months (180 days) after the final dose, she could be included in the study.
16. Patients who are determined to be inappropriate for participation in this study by the investigator or subinvestigator.

    [ACM regimen part] In addition to the exclusion criteria cfor all parts, patients who meet any one of the following criteria 17 to 21 will be excluded from the ACM regimen part.
17. Have the cumulative total exposure of anthracycline, daunorubicin-equivalent dose, exceeds 360 mg/m2 (body surface area) at entry.
18. Received other leukemia treatment within 21 days prior to entry.
19. Have a history of radiation therapy on the mediastinum.
20. Have sustained ≥ Grade 2 adverse drug reaction (except alopecia) as specified in CTCAE v4.03, which developed by the previous treatment.
21. Have a history of hypersensitivity against any one of cytarabine, mitoxantrone, or contained excipients.

    [A+7+3 regimen part] In addition to the exclusion criteria for all parts, patients who meet any one of the following criteria 22 to 23 will be excluded from the A+7+3 regimen part.
22. Have the cumulative total exposure of anthracycline, daunorubicin-equivalent dose, exceeds 100 mg/m2 (body surface area) at entry.
23. Have a history of hypersensitivity against any one of cytarabine, daunorubicin, or contained excipients.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability in Japanese AML patients by CTCAE v4.0 | 2 months
  Safety and tolerability of DSP-2033 (Alvocidib) in combination with cytarabine/mitoxantrone (ACM regimen) in Japanese patients with relapsed or refractory AML and in combination with cytarabine/daunorubicin (A+7+3 regimen) in Japanese newly diagnosed AML patients.
  Safety and tolerability analyses:The number of subjects with treatment-related adverse events as assessed by CTCAE v4.0. The number of subjects with DLT and incidence rate during the DLT evaluation period.

SECONDARY OUTCOMES:
To evaluate peak plasma concentration (Cmax) of ACM regimen and A+7+3 regimen in Japanese | 14 days
  Pharmacokinetics of individual drugs of ACM regimen in Japanese patients with relapsed or refractory AML and A+7+3 regimen in Japanese newly diagnosed AML patients.
  Pharmacokinetic analyses:Pharmacokinetic parameters of Maximum Plasma Concentration [Cmax] DSP-2033, DSP-2033 glucuronide (Alvo-G), cytarabine, mitoxantrone, and daunorubicin.
To evaluate Area under the plasma concentration versus time curve (AUC) of ACM regimen and A+7+3 regimen in Japanese | 14 days
  Pharmacokinetics of individual drugs of ACM regimen in Japanese patients with relapsed or refractory AML and A+7+3 regimen in Japanese newly diagnosed AML patients.
  Pharmacokinetic analyses:Pharmacokinetic parameters of Area Under the Curve [AUC] DSP-2033, DSP-2033 glucuronide (Alvo-G), cytarabine, mitoxantrone, and daunorubicin.
To evaluate the Anti-tumor effects based on bone-marrow blasts | 2 months
  * Complete remission rate (CR rate)
  * CR with incomplete hematologic recovery (CRi rate)
  * Combined Complete remission rate (CRc rate): a total of CR rate and CRi rate
  * Partial remission rate (PR rate)
  (Evaluated by 2017 European Leukemia Net AML efficacy assessment criteria)
Event-free survival (EFS) (ACM regimen part only) | 12 months
  EFS of ACM regimen in Japanese patients with relapsed or refractory AML.
Overall survival (OS) (ACM regimen part only) | 12 months
  OS of ACM regimen in Japanese patients with relapsed or refractory AML.

CONTACTS AND LOCATIONS:
Locations (11):
- Japan (11):
  - Fukui University Hospital, Yoshida-gun, Fukui
  - Chugoku Central Hospital, Fukuyama, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Tokai University Hospital, Isehara, Kanagawa
  - Osaka City Hospital Organization, Miyakojima-ku, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Fukushima Medical University Hospital, Fukushima

REFERENCES:
- [Derived] Ikezoe T, Ando K, Onozawa M, Yamane T, Hosono N, Morita Y, Kiguchi T, Iwasaki H, Miyamoto T, Matsubara K, Sugimoto S, Miyazaki Y, Kizaki M, Akashi K. Phase I study of alvocidib plus cytarabine/mitoxantrone or cytarabine/daunorubicin for acute myeloid leukemia in Japan. Cancer Sci. 2022 Dec;113(12):4258-4266. doi: 10.1111/cas.15458. Epub 2022 Oct 10. PMID 35689544